CLINICAL TRIAL: NCT06120465
Title: Yoga Outcomes Get Assessed in Cystic Fibrosis
Brief Title: YOGA-CF (Yoga Outcomes Get Assessed in Cystic Fibrosis)
Acronym: YOGA-CF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YOGA-CF
Record Dates: First submitted 2023-09-19; First posted 2023-11-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Cystic Fibrosis
Keywords: Yoga
MeSH Terms: conditions — Cystic Fibrosis | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga intervention group (Active Comparator): 12 week programme of yoga - encouraged to complete 1 live class and one pre-recorded class a week. Participants will continue with usual cystic fibrosis care.
  Interventions: Other: Yoga
- Control group (No Intervention): Usual cystic fibrosis care.

INTERVENTIONS:
Other: Yoga — Yoga classes
  Arms: Yoga intervention group

SUMMARY:
The goal of this clinical trial is to investigate the effects of yoga participation for adults with cystic fibrosis.

The main question it aims to answer is: does participation in yoga affect health-related quality of life for adults with cystic fibrosis?

Researchers will compare a group completing a 12-week yoga programme alongside usual cystic fibrosis care, to a group completing usual care alone to see if the addition of yoga effects health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of CF (confirmed by standard criteria; (Farrell et al. 2017))

Sixteen years of age or over

Home internet access

Ability to complete questionnaires in English

Stable CF disease as judged by the investigator, a senior CF clinician

Exclusion Criteria:

Inability to consent for treatment or measurement

Current participation in another interventional study of a medicinal product

Current haemoptysis (greater than streaking in the sputum)

Known pregnancy at time of recruitment

Forced expiratory volume in 1 second (FEV1) below 30% predicted at baseline

Use of ambulatory oxygen therapy, long-term oxygen therapy (LTOT) or non-invasive ventilation

Current regular participation in yoga practice

Current neurological or musculoskeletal injury which would prevent completion of yoga

Diagnosis of osteoporosis (bone density Z score <-2.5) or history of spontaneous spinal fractures

Uncontrolled gastroesophageal reflux

Acute pulmonary exacerbation within 28 days of screening

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory Health- related quality of life - measured by the respiratory domain of the Cystic Fibrosis Questionnaire - Revised. | Baseline, 12 and 24-weeks
  Cystic Fibrosis Questionnaire - Revised (CFQ-R) respiratory domain.Scores range from 0 to 100, with higher scores indicating better health.

SECONDARY OUTCOMES:
Other Health-related quality of life domains - captured on the Cystic Fibrosis Questionnaire - Revised (CFQ-R) | Baseline, 12 and 24-weeks
  Cystic Fibrosis Questionnaire - Revised (CFQ-R) other eleven domains. Scores range from 0 to 100, with higher scores indicating better health.
One Minute Sit to Stand Test | Baseline, 12 and 24-weeks
  Participant stands up and sits down from a chair for one minute and the number of completed sit-to-stands is recorded.
Forced Expiratory Volume in 1 second | Baseline, 12 and 24-weeks
  Forced expiratory volume in 1 second (FEV1) obtained through spirometry. Measured in litres and percentage predicted (using Global Lung Index equations)
Forced vital capacity (FVC) | Baseline, 12 and 24-weeks
  Forced vital capacity obtained through spirometry. Measured in litres and percentage predicted (using Global Lung Index equations)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Simmonds, Principal Investigator — Royal Brompton Hospital, Guys and St Thomas's Foundation Trust
Locations (1):
- The Royal Brompton Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stanford GE, Scarborough P, Charman SC, Cameron RA, Wagner AP, Simmonds NJ. Yoga Outcomes Get Assessed in Cystic Fibrosis (YOGA-CF): protocol of a multicentre interventional randomised controlled clinical trial-investigating effects of a 12-week yoga intervention for adults with cystic fibrosis. BMJ Open Respir Res. 2026 Jan 6;13(1):e003405. doi: 10.1136/bmjresp-2025-003405. PMID 41494700